CLINICAL TRIAL: NCT02150317
Title: A Prospective Randomized Trial Comparing Transcatheter Arterial Chemoembolization (TACE) Followed by Sorafenib Versus TACE Alone for Advanced Hepatocellular Carcinoma
Brief Title: Transarterial Chemoembolization (TACE) Plus Sorafenib Versus TACE for Advanced Hepatocellular Carcinoma
Acronym: TACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2013-001-08
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Carcinoma, Hepatocellular; Chemoembolization, Therapeutic; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE+Sorafenib (Active Comparator): TACE followed by Sorafenib
  Interventions: Procedure: TACE+Sorafenib
- TACE (Experimental): TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE+Sorafenib — TACE followed by Sorafenib
  Other Names: TACE followed by Sorafenib
  Arms: TACE+Sorafenib
Procedure: TACE — TACE alone
  Arms: TACE

SUMMARY:
The aim of this study is to compare the outcomes of Transarterial Chemoembolization (TACE) followed by Sorafenib with TACE alone in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* at least 2 radiologic imaging showing characteristic features of hepatocellular carcinoma or cytologic/histologic evidence.
* tumor in liver and radiologically definable vascular invasion or extrahepatic metastasis.
* Criteria of liver function: Child A-B level, serum bilirubin ≤ 1.5 times the upper limit of normal value,alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
* No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal.
* Hb ≥90g/L,white blood cell count ≥3.000 cells/mm³,platelets ≥80.000 cells/mm³
* Patients who can understand this trial and have signed information consent

Exclusion Criteria:

* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer.
* Patients with other diseases which may affect the treatment mentioned.
* Patients with a medical history of other malignant tumors.
* Subjects participating in other clinical trials.
* liver function:Child C.
* no pathological evidence of hepatocellular carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the overall survival rate of each group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ai-jun Li, M.D., Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China